CLINICAL TRIAL: NCT06606587
Title: Evaluation of the Effectiveness of the Comfort-In Needle-Free Injector System During Palatal Infiltrative Anesthesia in Children
Brief Title: Effectiveness of the Comfort-In Needle Free Injection System During Palatal Infiltrative Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Halenur Altan, Associated professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NecmettinEU02
Record Dates: First submitted 2024-08-15; First posted 2024-09-23 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-05

CONDITIONS: Physiological Effects of Drugs; Anesthetics
Keywords: needle-free injection; palatal injection; pain; procedural pain
MeSH Terms: conditions — Pain; Pain, Procedural

STUDY DESIGN:
Intervention Model Description: The method to be applied to patients who met the inclusion criteria was determined randomly with the help of a computer.
Masking Description: When giving data to the statistician, he will not be told which group the data is in. The data will be changed to a and b to try to prevent bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group Experimental: Application of Comfort-in Jet Injection Method (Experimental): Application of Comfort-in Jet Injection Method Comfort-in jet injection method was used for palatal anesthesia of the permanent 1st molar. Using a silicone flat cap, it was placed 5 mm below the palatal gingival margin, close to the free gingiva, and with a steep angle. 0.3 ml of anesthetic solution was administered by pressing the jet injection system button. 1 mL Articaine Hydrochloride (Ultracaine D-S forte, Hoechst, Canada) containing 1/100,000 epinephrine was used as a local anesthetic agent in the injections. 31 patients were included in this group and the procedure was performed. After waiting for 2 minutes, the anesthetized area was probed with the help of a probe (probing gingiva) to check whether the anesthesia had taken effect. Afterwards, buccal infiltration anesthesia was performed with the help of a traditional dental injector and tooth extraction was performed.
  Interventions: Device: Comfort-in Jet Injection Method
- Group Control: Application of Traditional Dental Injection Method (Other): Application of Traditional Dental Injection Method Palatal injection; It was applied 5-10 mm below the palatal gingival margin*, on the attached gum, and with a 45-degree needle angle. After needle entry, 0.2-0.3 mL of anesthetic solution was stored when bone contact was removed (3-5 mm). 1 mL Articaine Hydrochloride (Ultracaine D-S forte, Hoechst, Canada) containing 1/100,000 epinephrine and a 27 G dental needle were used as local anesthetic agents for injections. 25 patients were included in this group and the procedure was performed. After waiting for 5 minutes, the anesthetized area was probed with the help of a probe (probing gingiva) to check whether the anesthesia had taken effect. Afterwards, buccal infiltration anesthesia was performed with the help of a traditional dental injector and tooth extraction was performed.
  Interventions: Other: Traditional Dental Injection

INTERVENTIONS:
Device: Comfort-in Jet Injection Method — Application of Comfort-in Jet Injection Method: Comfort-in jet injection method was used for palatal anesthesia of the permanent 1st molar.
  Arms: Group Experimental: Application of Comfort-in Jet Injection Method
Other: Traditional Dental Injection — Application of Traditional Dental Injection Method: Traditional Dental Injection method was used for palatal anesthesia of the permanent 1st molar.
  Arms: Group Control: Application of Traditional Dental Injection Method

SUMMARY:
The goal of this randomized clinical trial is to compare two different injection methods in children. The main question it aims to answer is:

Is the needle-free injection method more painless than the traditional dental method?

Two different methods will be used for children to perform anesthesia for extraction permanent molars.

DETAILED DESCRIPTION:
Study Groups and Study Design: 56 volunteer children between the ages of 6-15 who applied to Faculty of Dentistry Department of Pedodontics clinic with their parents were included in our study. Volunteer children with an indication for maxillary permanent first molar tooth extraction were randomly divided into two groups and included in the study. For randomization, methods were written on two different envelopes and the child was allowed to choose the envelope. The child was assigned to the selected method. Group Control: Application of Traditional Dental Injection Method Palatal injection; It was applied 5-10 mm below the palatal gingival margin*, on the attached gum, and with a 45-degree needle angle. After needle entry, 0.2-0.3 mL of anesthetic solution was stored when bone contact was removed (3-5 mm). 1 mL Articaine Hydrochloride (Ultracaine D-S forte, Hoechst, Canada) containing 1/100,000 epinephrine and a 27 G dental needle were used as local anesthetic agents for injections. 25 patients were included in this group and the procedure was performed. After waiting for 5 minutes, the anesthetized area was probed with the help of a probe (probing gingiva) to check whether the anesthesia had taken effect. Afterwards, buccal infiltration anesthesia was performed with the help of a traditional dental injector and tooth extraction was performed. Group Experimental: Application of Comfort-in Jet Injection Method Comfort-in jet injection method was used for palatal anesthesia of the permanent 1st molar. Using a silicone flat cap, it was placed 5 mm below the palatal gingival margin, close to the free gingiva, and with a steep angle. 0.3 ml of anesthetic solution was administered by pressing the jet injection system button. 1 mL Articaine Hydrochloride (Ultracaine D-S forte, Hoechst, Canada) containing 1/100,000 epinephrine was used as a local anesthetic agent in the injections. 31 patients were included in this group and the procedure was performed. After waiting for 2 minutes, the anesthetized area was probed with the help of a probe (probing gingiva) to check whether the anesthesia had taken effect. Afterwards, buccal infiltration anesthesia was performed with the help of a traditional dental injector and tooth extraction was performed.

ELIGIBILITY:
Inclusion Criteria:

Child patient between the ages of 6-16, Requiring extraction of maxillary permanent molars and premolars with bilateral palatal infiltration anesthesia, Showing "positive" and "definitely positive" behavior during examination according to the Frankl scale, Family volunteers, No medical or developmental disease

Exclusion Criteria:

If there are medical or developmental disorders, If there is a chronic disease, If there is an allergy to anesthetic solutions, If there is any pathology in the anesthesia area, If the Frankl scale is "negative" and "definitely negative", If the mouth opening is not sufficient, If there is no need for symmetrical treatment in the teeth

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Pain Perception of Wong-Baker Scale | After the anesthesia method is applied, the patient is asked to score the pain they feel
  The investigators expect the comfort-in jet injection method to produce a lower score on the Wong-Baker pain scale than the traditional anesthesia method.The Wong-Baker pain scale is scored between 0-10. 0 means the patient has no pain and 10 means they feel very severe pain.
Pain Perception of The Face, Legs, Activity, Cry, and Consolability (FLACC) scale | The video taken to look at the patients body reactions during the application of the anesthesia method is evaluated and scored after the procedure is completed.
  The investigators expect the comfort-in jet injection method to produce a lower score on the FLACC scale applied to pain acceptance in pediatric patients compared to the traditional anesthesia method. The FLACC pain scale is scored between 0-10. 0 means that the patients pain acceptance is good and 10 means that the pain acceptance is low.

CONTACTS AND LOCATIONS:
Overall Officials: Halenur Altan, Study Chair — Necmetttin Erbakan University Dentistry Faculty
Locations (1):
- : Halenur Altan, assoc. prof., Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Altan H, Belevcikli M, Cosgun A, Demir O. Comparative evaluation of pain perception with a new needle-free system and dental needle method in children: a randomized clinical trial. BMC Anesthesiol. 2021 Dec 1;21(1):301. doi: 10.1186/s12871-021-01524-1. PMID 34852779